CLINICAL TRIAL: NCT05027269
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1/2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple-Doses of AOC 1001 Administered Intravenously to Adult Myotonic Dystrophy Type 1 (DM1) Patients
Brief Title: Study of AOC 1001 in Adult Myotonic Dystrophy Type 1 (DM1) Patients
Acronym: MARINA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Avidity Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AOC 1001-CS1
Record Dates: First submitted 2021-08-24; First posted 2021-08-30 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: DM1; Myotonic Dystrophy 1; Myotonic Dystrophy; Myotonic Dystrophy Type 1 (DM1); Dystrophy Myotonic; Myotonic Disorders; Steinert Disease; Myotonic Muscular Dystrophy
Keywords: DM1; Myotonic Dystrophy 1; Myotonic Dystrophy Type 1 (DM1); Myotonic Dystrophy; DM; Dystrophy Myotonic; Myotonic Disorders; Steinert Disease; MARINA; Avidity Biosciences; Avidity; AOC 1001; Myotonic Muscular Dystrophy
MeSH Terms: conditions — Myotonic Dystrophy; Myotonic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A Single Dose: AOC 1001 Dose Level 1 (Experimental): AOC 1001 will be administered once.
  Interventions: Drug: AOC 1001
- Part A Single Dose: Placebo (Placebo Comparator): Saline will be administered once.
  Interventions: Drug: Placebo
- Part B Multiple Ascending Dose: AOC 1001 Dose Levels 2 & 3 (Experimental): AOC 1001 will be administered three times.
  Interventions: Drug: AOC 1001
- Part B Multiple Ascending Dose: Placebo (Placebo Comparator): Saline will be administered three times.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AOC 1001 — AOC 1001 will be administered by intravenous (IV) infusion.
  Arms: Part A Single Dose: AOC 1001 Dose Level 1; Part B Multiple Ascending Dose: AOC 1001 Dose Levels 2 & 3
Drug: Placebo — Placebo will be administered by intravenous (IV) infusion.
  Arms: Part A Single Dose: Placebo; Part B Multiple Ascending Dose: Placebo

SUMMARY:
AOC 1001-CS1 is a randomized, double-blind, placebo-controlled, Phase 1/2 study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single and multiple-doses of AOC 1001 Administered Intravenously to Adult Myotonic Dystrophy Type 1 (DM1) patients (MARINA).

Part A is a single dose design with 1 cohort (dose level). In Part A, the patient duration is 6 months as the treatment period is 1 day followed by a 6 month follow-up period.

Part B is a multiple-ascending dose design with 2 cohorts (dose levels). In Part B, the patient duration is 6 months as the treatment period is 3 months followed by a 3 month follow-up period.

ELIGIBILITY:
Key Inclusion Criteria:

* Genetic diagnosis of DM1 (CTG repeat length ≥ 100)
* Clinician assessed signs of DM1
* Ability to walk independently (orthoses and ankle braces allowed) for at least 10 meters at screening

Key Exclusion Criteria:

* Diabetes that is not adequately controlled
* BMI > 35 kg/m2
* Uncontrolled hypertension
* Congenital DM1
* History of tibialis anterior (TA) biopsy within 3 months of Day 1 or planning to undergo TA biopsies during study period
* Recently treated with an investigational drug
* Treatment with anti-myotonic medication within 14 days of Day 1

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Frequency of treatment emergent adverse events (TEAEs) | Through study completion, up to Day 183

SECONDARY OUTCOMES:
Plasma pharmacokinetic (PK) parameters | Through study completion, up to Day 183
  Maximum plasma concentration (Cmax)
Plasma pharmacokinetic (PK) parameters | Through study completion, up to Day 183
  Time to maximum plasma concentration (Tmax)
Plasma pharmacokinetic (PK) parameters | Through study completion, up to Day 183
  Terminal Half-life (t1/2)
Plasma pharmacokinetic (PK) parameters | Through study completion, up to Day 183
  Area Under the Concentration-time Curve (AUC)
Urine pharmacokinetic (PK) parameters | Through study completion, up to Day 183
  fraction excreted (fe) in urine
AOC 1001 levels in muscle tissue | Through study completion, up to Day 183
Change and percentage change from baseline in DMPK mRNA knockdown | Through study completion, up to Day 183
Change and percentage change from baseline in Spliceopathy | Through study completion, up to Day 183

CONTACTS AND LOCATIONS:
Overall Officials: Li Tai, MD, Study Director — Avidity Biosciences, Inc.
Locations (8):
- United States (8):
  - University of California Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of Colorado, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Rochester Medical Center, Rochester, New York
  - Ohio State University, Columbus, Ohio
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.aviditybiosciences.com/